CLINICAL TRIAL: NCT01440855
Title: Efficacy and Feasibility of a Psychosocial Intervention Within CCOP Context: Evaluation of the Facing Forward Guide to Facilitate Life After Active Cancer Treatment (CCOP:Community Clinical Oncology Program)
Brief Title: Evaluation of the Efficacy of National Cancer Institute's Facing Forward Booklet in the Cancer Community Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB06803; U10CA101178-03 (NIH)
Record Dates: First submitted 2011-09-22; First posted 2011-09-27 (Estimated); Last update posted 2011-10-04 (Estimated); Status verified 2011-09

CONDITIONS: Prostate Cancer; Breast Cancer; Colorectal Cancer; Thoracic Cancer
Keywords: Survivorship; cancer control; psychosocial interventions; Facing Forward
MeSH Terms: conditions — Prostatic Neoplasms; Breast Neoplasms; Colorectal Neoplasms | interventions — cytokine inducible SH2-containing protein

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CIS Fact Sheet (CIS: Cancer Information Service) (Active Comparator): CIS Fact Sheet, available on the Cancer Information Service website. Used to control for attention. 5-page document provides information about the CIS:What is it, How can CIS information specialists help me, How can I use CIS's services. Also includes definitions of glossary terms and a table of email and website addresses.
  Interventions: Other: CIS (Cancer Information Service) Information Sheet
- Facing Forward booklet (Experimental): NCI's Facing Forward 61-page booklet, which describes common feelings and reactions that cancer survivors experience during the re-entry phase and offers behavioral recommendations to help them through this period, i.e., ways of dealing with common problems and guidelines for managing physical, social, and emotional health. Booklet sections: Congratulations on Finishing Your Cancer Treatment, Getting Follow-up Medical Care, Ways to Manage Physical Changes, Body Changes and Intimacy, Your Feelings, Social and Work Relationships, Reflection, 6-page Appendix, which provides information on Financial and Legal Matters, and Resource Organizations.
  Interventions: Other: Facing Forward booklet

INTERVENTIONS:
Other: CIS (Cancer Information Service) Information Sheet — CIS Fact Sheet, available on the Cancer Information Service website. Used to control for attention. 5-page document provides information about the CIS:What is it, How can CIS information specialists help me, How can I use CIS's services. Also includes definitions of glossary terms and a table of email and website addresses.
  Arms: CIS Fact Sheet (CIS: Cancer Information Service)
Other: Facing Forward booklet — NCI's (NCI: National Cancer Institute) Facing Forward 61-page booklet, which describes common feelings and reactions that cancer survivors experience during the re-entry phase and offers behavioral recommendations to help them through this period, i.e., ways of dealing with common problems and guidelines for managing physical, social, and emotional health. Booklet sections: Congratulations on Finishing Your Cancer Treatment, Getting Follow-up Medical Care, Ways to Manage Physical Changes, Body Changes and Intimacy, Your Feelings, Social and Work Relationships, Reflection, 6-page Appendix, which provides information on Financial and Legal Matters, and Resource Organizations.
  Arms: Facing Forward booklet

SUMMARY:
This study was designed to provide a preliminary evaluation of the efficacy and usability of the 2004 revised version of the booklet, Facing Forward , Life After Cancer Treatment, (hereafter,Facing Forward) published by the National Cancer Institute. Facing Forward provides early stage cancer patients during the period after completing active treatment practical ways of dealing with common problems, including guidelines for managing physical, social, and emotional health. Assessments were completed at the patient's final cancer treatment visit. Follow-up assessments occurred eight weeks and 6 months later. The initial assessments covered background information (demographics, medical status), use of educational materials, survivorship activities, and psychological factors. The follow-up assessments included use of actions recommended in Facing Forward, ratings of Facing Forward with respect the booklet's informativeness, helpfulness, understandability, and extent read, the same psychological measures used initially, and a measure of self-efficacy.

DETAILED DESCRIPTION:
This study was designed to provide a preliminary evaluation of the efficacy and usability of the 2004 revised version of the booklet, Facing Forward, Life After Cancer Treatment (hereafter,Facing Forward)published by the National Cancer Institute. Facing Forward provides early stage cancer patients during the period after completing active treatment practical ways of dealing with common problems, including guidelines for managing physical, social, and emotional health. The study employed a randomized controlled repeated measures design and compared Facing Forward with a control document published by the National Cancer Institute, The Cancer Information Service: Questions and Answers. The intervention arm received both Facing Forward and the control document and the control arm received only the latter. Assessments were completed at baseline, which occurred at the patient's final cancer treatment visit or alternatively at the first follow-up visit for those scheduled to be evaluated and/or restaged within 28 days of their last treatment visit. The first follow-up assessment occurred eight weeks following the baseline assessment via mail-home materials, and the second occurred 6 months following the baseline assessment, again via mail-home materials. Baseline measures included background information (demographics, medical status), use of educational materials, survivorship activities engaged in, and psychological factors. The 8-week and 6-month assessments included uptake of actions recommended in Facing Forward, and ratings of Facing Forward with respect to its usability, including the booklet's informativeness, helpfulness, understandability, and extent read, and the same psychological factors assessed at baseline.

ELIGIBILITY:
Inclusion Criteria:

* current age at or above 18 years;
* breast, colorectal, prostate, and/or thoracic cancer diagnosis,stage I, II, IIIa;
* approaching or attending the last treatment appointment of chemotherapy and or radiation therapy for the cancer diagnosis
* English speaking (able to read English at an 8th grade level);
* have a mailing address;
* have residential phone service;
* able to give informed consent.

Exclusion Criteria:

* patients who have received surgery only with no adjuvant therapy;
* second primary cancer or recurrent disease;
* patients receiving brachytherapy only

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2005-02; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Reported uptake of behavioral actions recommended in Facing Forward | Baseline
  Items asked whether the respondent engaged in each recommended behavior (Yes or No); affirmative responses to the items comprising each subscale were summed to create four subscale scores:use of follow-up medical care (6 items; e.g., have you developed a wellness plan?), management of side effects of management (7 items; e.g., have you used any tips for regaining your appetite? ), uptake of stress management (8 items; e.g., have you used relaxation techniques? ), management of social and financial matters management (7 items; e.g., have you used suggested tips for dealing with family issues?.
Reported uptake of behavioral actions recommended in Facing Forward | 8-weeks post-baseline
  Items asked whether the respondent engaged in each recommended behavior (Yes or No); affirmative responses to the items comprising each subscale were summed to create four subscale scores:use of follow-up medical care (6 items; e.g., have you developed a wellness plan?), management of side effects of management (7 items; e.g., have you used any tips for regaining your appetite? ), uptake of stress management (8 items; e.g., have you used relaxation techniques? ), management of social and financial matters management (7 items; e.g., have you used suggested tips for dealing with family issues?.
Reported uptake of behavioral actions recommended in Facing Forward | 6-months post-baseline
  Items asked whether the respondent engaged in each recommended behavior (Yes or No); affirmative responses to the items comprising each subscale were summed to create four subscale scores:use of follow-up medical care (6 items; e.g., have you developed a wellness plan?), management of side effects of management (7 items; e.g., have you used any tips for regaining your appetite? ), uptake of stress management (8 items; e.g., have you used relaxation techniques? ), management of social and financial matters management (7 items; e.g., have you used suggested tips for dealing with family issues?.

SECONDARY OUTCOMES:
Usability of Facing Forward | Eight weeks post-baseline
  Informativeness of booklet with respect to post-treatment challenges (8 items);confidence about the participant's ability to deal with each of the challenges (8 items);helpfulness (15 items)and understandability (15 items)of booklet as a whole and of 6 booklet sections and 3 appendices; likelihood of uptake(16 items)of engaging in behaviors recommended in booklet;whether (9 items) and extent to which (9 items)6 booklet sections and 3 appendices was read.
Usability of Facing Forward | 6 months post-baseline
  Informativeness of booklet with respect to post-treatment challenges (8 items);confidence about the participant's ability to deal with each of the challenges (8 items);helpfulness (15 items)and understandability (15 items)of booklet as a whole and of 6 booklet sections and 3 appendices; likelihood of uptake(16 items)of engaging in behaviors recommended in booklet;whether (9 items) and extent to which (9 items)6 booklet sections and 3 appendices was read.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne M Miller-Halegoua, PhD, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States